CLINICAL TRIAL: NCT02686385
Title: Efficacy of N-acetylcysteine With or Without Steroids in Drug Induced Liver Injury: A Prospective Randomized Controlled Trial
Brief Title: Efficacy of N-acetylcysteine With or Without Steroids in Drug Induced Liver Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Steroids were given for 2 patients who had biopsy proven Drug induced Liver Injury and both have them developed sepsis.
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-DILI-001
Record Dates: First submitted 2016-02-08; First posted 2016-02-19 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2016-08

CONDITIONS: Drug Induced Liver Injury
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury | interventions — Prednisolone; Acetylcysteine

ARMS (2):
- Prednisolone + N-Acetylcysteine (Experimental): Prednisolone for 20 days with NAC (N-Acetylcysteine) NAC (N-Acetylcysteine) dosing-Loading dose: 150 mg/kg IV; mix in 200 mL of 5% dextrose in water (D5W) and infuse over 1 h Dose 2: 50 mg/kg IV in 500 mL D5W over 4 h Dose 3: 100 mg/kg IV in 1000 mL D5W over 16 h
  Interventions: Drug: Prednisolone; Drug: N-Acetylcysteine
- N-Acetylcysteine (Active Comparator): NAC (N-Acetylcysteine) dosing-Loading dose: 150 mg/kg IV; mix in 200 mL of 5% dextrose in water (D5W) and infuse over 1 h Dose 2: 50 mg/kg IV in 500 mL D5W over 4 h Dose 3: 100 mg/kg IV in 1000 mL D5W over 16 h
  Interventions: Drug: N-Acetylcysteine

INTERVENTIONS:
Drug: Prednisolone
  Arms: Prednisolone + N-Acetylcysteine
Drug: N-Acetylcysteine — NAC (N-Acetylcysteine) dosing-Loading dose: 150 mg/kg IV; mix in 200 mL of 5% dextrose in water (D5W) and infuse over 1 h Dose 2: 50 mg/kg IV in 500 mL D5W over 4 h Dose 3: 100 mg/kg IV in 1000 mL D5W over 16 h

SUMMARY:
Intervention - Subjects will be randomized to 2 groups

Group A - subjects will receive Prednisolone for 20 days with NAC (N-Acetylcysteine)

Group B - will receive NAC (N-Acetylcysteine) only NAC (N-acetylcysteine) dosing

Loading dose: 150 mg/kg IV; mix in 200 mL of 5% dextrose in water (D5W) and infuse over 1 hour

Dose 2: 50 mg/kg IV in 500 mL D5W over 4 h

Dose 3: 100 mg/kg IV in 1000 mL D5W over 16 h

* Monitoring and assessment-Liver Biopsy at baseline and at 3 months, Liver Function Test at regular intervals.
* Stopping rule-Development of sepsis, worsening of Liver functions.

ELIGIBILITY:
Inclusion Criteria:

* All patients with severe DILI (Drug Induced Liver Injury)
* Age more than or equal to 18 years

Exclusion Criteria:

* Patients with HAV (Hepatitis A Virus), HBV (Hepatitis B Virus), HCV (Hepatitis C Virus), HEV (Hepatitis E Virus) Positive
* Patients with sepsis
* AMA positive
* Low Ceruloplasmin
* Transferrin saturation >45%
* Patients with Cirrhosis
* Patients with h/o jaundice prior to the intake of drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with normalization of LFT (Liver Function Test) in both groups. | 20 days
  Normalization of LFT (Liver Function Test) which is defined as Total bilirubin within normal limits.

SECONDARY OUTCOMES:
Improvement in of Histology. | 20 days
  Improvement is defined as decrease in inflammation, decrease in cholestasis.
Improvement in CBC profile | 20 days
  Improvement is defined normalization of CBC profile.
Improvement in coagulation profile | 20 days
  Improvement is defined normalization of Coagulation profile.
Improvement in KFT profile | 20 days
  Improvement is defined normalization of KFT profile.
Proportion of patients develop adverse effects in both groups. | 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr Anand Kulkarni V, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India